CLINICAL TRIAL: NCT01980173
Title: Medico-economic Comparison of Postpartum Hemorrhage Management Using the Bakri Balloon and Standard Care
Acronym: Bakri
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2012/VL-04; 2013-A00914-41 (Other: RCB number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-08 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2016-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Bakri balloon
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Bakri balloon (Experimental): Patients randomized to this arm will be treated using the Bakri balloon.
  Intervention: Bakri balloon
  Interventions: Device: Bakri balloon
- Without Bakri balloon (Active Comparator): Patients randomized to this arm will receive routine care not including the Bakri Balloon.
  Intervention: Routine Care
  Interventions: Procedure: Routine care

INTERVENTIONS:
Procedure: Routine care — Following diagnosis with post-partum hemorrhage, an initial 30 minute phase corresponding to current recommendations, an injection of sulprostone, a demonstrated inefficacy of sulprostone 20 minutes after the injection and finally randomization, patients in this arm of the study will continue to have routine care.
  Arms: Without Bakri balloon
Device: Bakri balloon — Following diagnosis with post-partum hemorrhage, an initial 30 minute phase corresponding to current recommendations, an injection of sulprostone, a demonstrated inefficacy of sulprostone 20 minutes after the injection and finally randomization, patients in this arm will be treated with the immediate placement of a Bakri balloon, followed by routine care if necessary.
  Arms: With Bakri balloon

SUMMARY:
This study concerns women diagnosed with postpartum hemorrhage and requiring sulprostone therapy. Included patients are randomized to two arms: the "Sulprostone + Bakri balloon" arm versus the "Sulprostone alone" arm.

The main objective of this study is to compare the efficiency of a care strategy including the Bakri balloon to that of routine care without the Bakri balloon via a cost-consequence study juxtaposing costs and the necessity of invasive procedures (arterial embolization, ligation of arteries, hysterectomy, intrauterine sutures) for controlling postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* The patient, her person-of-trust, must have given his/her consent and signed the consent form / inclusion decision made by the investigator when a person-of-trust is absent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is able to fluently read and speak French
* Blood loss > 500ml and sulprostone treatment is insufficient at 20 minutes
* Duration of pregnancy > 32 weeks of amenorrhea
* Uterine atony

Exclusion Criteria:

* The patient is participating in another study except for the followin studies: ElastoMAP, ElastoDéclench, Papillo PMA, GrossPath, LXRs, DGPostPartum
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient cannot read French
* The patient was transferred to another center not among the centers participating in this study
* The patient has a contraindication for a treatment used in this study (Sulprostone), or an incompatible treatment combination
* The patient has a contraindication for third level techniques
* The patient has at least one of the following conditions: chorioamnionitis, cervical cancer, uterine rupture, anatomical abnormality preventing the introduction of the device, purulent infection of the vagina, cervix or uterus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
The % of patients requiring invasive measures for postpartum hemorrhage control. | Hospital stay (expected max of 15 days).
The total cost (€) associated with the postpartum hemorrhage management strategy. | Hospital stay (expected max of 15 days).

SECONDARY OUTCOMES:
The delay required to stop bleeding post-delivery (min) | post-partum (expected maximum of a few hours)
The delay required to stop bleeding post-diagnosis (min) | post-partum (expected maximum of a few hours)
The percentage of patients still bleeding 30 minutes after sulprostone injection | 30 minutes after sulprostone injection (day 0)
Blood loss (ml) 30 minutes after diagnosis | 30 minutes after diagnosis (day 0)
Blood loss (ml) 1 hour after diagnosis | 1 hour after diagnosis (day 0)
Blood loss (ml) 2 hours after diagnosis | 2 hours after diagnosis (day 0)
Blood loss (ml) 24 hours after diagnosis | 24 hours after diagnosis (day 1)
Blood pressure | Upon diagnosis (day 0)
Blood pressure | 30 minutes after diagnosis (day 0)
Blood pressure | 120 minutes after diagnosis (day 0)
Blood pressure | 24 hours after diagnosis (day 1)
Blood pressure | upon sulprostone injection (day 0)
Blood pressure | when placing the Bakri balloon (day 0)
Blood pressure | when performing invasive techniques (expected day 0 or 1)
Heart rate | Upon diagnosis (day 0)
Heart rate | 30 minutes after diagnosis (day 0)
Heart rate | 120 minutes after diagnosis (day 0)
Heart rate | 24 hours after diagnosis (day 1)
Heart rate | upon sulprostone injection (day 0)
Heart rate | when placing the Bakri balloon (day 0)
Heart rate | when performing invasive techniques (expected day 0 or 1)
The % of patients requiring blood transfusion. | Hospital stay (expected max of 15 days).
The % of patients requiring intravenous iron. | Hospital stay (expected max of 15 days).
The quantity of packed red cells, platelet concentrate and fresh frozen plasma consumed | Hospital stay (expected max of 15 days).
Fibrinogen (g / l) | Upon diagnosis (day 0)
Fibrinogen (g / l) | Day 1
Fibrinogen (g / l) | Day 3
Hematocrit (%) | Upon diagnosis (day 0)
Hematocrit (%) | Day 1
Hematocrit (%) | Day 3
Hematocrit (%) | the month preceding delivery
Hemoglobin (g/dl) | Upon diagnosis (day 0)
Hemoglobin (g/dl) | Day 1
Hemoglobin (g/dl) | Day 3
Hemoglobin (g/dl) | the month preceding delivery
Prothrombin (%) | the month preceding delivery
Prothrombin (%) | Upon diagnosis (day 0)
Prothrombin (%) | Day 1
Prothrombin (%) | Day 3
Activated partial thromboplastin time (s) | the month preceding delivery
Activated partial thromboplastin time (s) | Upon diagnosis (day 0)
Activated partial thromboplastin time (s) | Day 1
Activated partial thromboplastin time (s) | Day 2
Length of hospital stay (days) | Expected max of 15 days
Length of ICU stay | expected max of 15 days
Antimullerian hormone level | Upon diagnosis (Day 0)
Antimullerian hormone level | 2 months after restart of menses
Amenorrhea at 3 months? yes/no | 3 months
  (Excluding breastfeeding women)
The presence of adhesions detected at hysteroscopy | 3 months after delivery if menses have restarted, or 2 months after the restart of menses (maximum of 1 year after inclusion)
pain will be assessed in both arms via a visual analog scale, duration, location, and use of analgesics | Day 1
pain will be assessed in both arms via a visual analog scale, duration, location, and use of analgesics | Day 3
temperature (°C) | Daily while in hospital (expected maximum of 15 days)
FSFI questionnaire (Female Sexual Function Index) | 6 months
Doppler ultrasound: intrauterine pressure | when placing the Bakri balloon; day 0
Doppler ultrasound: thickness of the uterine wall | when placing the Bakri balloon; day 0
Doppler ultrasound: inversed diastolic flow | when placing the Bakri balloon; day 0
Doppler ultrasound: intraluminal pressure | when placing the Bakri balloon; day 0
Doppler ultrasound: uterine artery perfusion pressure | when placing the Bakri balloon; day 0
Doppler ultrasound: uterine artery pulsatility index | when placing the Bakri balloon; day 0
IES-R scale (symptoms of post-traumatic stress) | 6 months
Vascular filling required? yes/no | Day 0
If vascular filling is required, volume and type of solution used. | Day 0
Were amines required? yes/no | Day 0

OTHER OUTCOMES:
Prophylactic antibiotherapy? yes/no | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (7):
- France (7):
  - CHU d'Angers - Hôtel-Dieu, Angers
  - APHP - Hôpital Antoine Beclere, Clamart
  - APHP - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - APHM - Hôpital Nord, Marseille
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374